CLINICAL TRIAL: NCT06623981
Title: Testing the Effectiveness and Implementation of an Evidence-Based Maternal Depression Treatment in an Urban Pediatric Asthma Clinic
Brief Title: The Exhale Study: Treating Maternal Depression in an Urban Pediatric Asthma Clinic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001112; K01MD018636 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-10-02 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Asthma in Children; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced IPT-B (Experimental): Enhanced Brief Interpersonal Psychotherapy
  Interventions: Behavioral: Enhanced Brief Interpersonal Psychotherapy
- Supplemented Usual Care (Active Comparator): Short-term care coordination
  Interventions: Behavioral: Supplemented Usual Care

INTERVENTIONS:
Behavioral: Enhanced Brief Interpersonal Psychotherapy — Enhanced IPT-B consists of a single, 45-60-minute pre-treatment engagement session followed by eight weekly, 45-minute individual sessions carried out within an 8-12-week timeframe.
  Arms: Enhanced IPT-B
Behavioral: Supplemented Usual Care — Usual care for caregivers with depressive symptoms involves the asthma clinic physician discussing the PHQ-9 results with the caregiver, providing brief psychoeducation on depression and giving the caregiver a written list of mental health resources. Usual care will be supplemented by providing short-term care coordination. Care coordination will involve assisting the participant in calling a mental health clinic to make an appointment and one follow-up phone call within two weeks.
  Arms: Supplemented Usual Care

SUMMARY:
The goal of this clinical trial is to test the effectiveness and implementation of delivering Enhanced Brief Interpersonal Psychotherapy (IPT-B), an evidence-based maternal depression treatment, to mothers of children under the age of 18 in an urban pediatric asthma clinic. Researchers will compare Enhanced IPT-B and supplemented usual care (brief care coordination). The main questions the trial aims to answer are:

1. Does Enhanced IPT-B decrease maternal depressive symptoms?
2. Does Enhanced IPT-B improve child asthma management and health outcomes (exacerbations, symptoms, control)?
3. What are the preliminary implementation outcomes of delivering Enhanced IPT-B in an urban pediatric asthma clinic?

DETAILED DESCRIPTION:
The purpose of the study is to determine the effectiveness and implementation of Brief Enhanced Interpersonal Psychotherapy (IPT-B), an evidence-based treatment for maternal depression, delivered in an urban pediatric asthma clinic. This study is a pilot Hybrid Type 1 Effectiveness-Implementation, single-blinded, prospective randomized controlled trial. A parallel two-group design will be used to evaluate the impact of the intervention (Enhanced IPT-B) among a sample of 48 Black mothers of children under the age of 18 with asthma. Mothers with PHQ-9 ≥ 8 will be identified in the asthma clinic through routine depression screening during the child's visit and recruited to participate in the study if they meet eligibility criteria. Following the informed consent process, mothers randomized to the intervention group will receive Enhanced IPT-B. Enhanced IPT-B consists of a single, 45-60-minute pre-treatment engagement session followed by eight weekly, 45-minute individual psychotherapy sessions carried out by a licensed mental health clinician within an 8-12-week timeframe. Mothers randomized to the comparison group will receive Supplemented Usual Care which involves short-term care coordination to access community mental health resources. Data on maternal mental health, child asthma management and outcomes, and child mental health will be collected from mothers and children at baseline, 3 months post-baseline, and 6 months post-baseline. Data on implementation outcomes will be collected from mothers and asthma clinic leadership and staff. Quantitative and qualitative data analysis strategies will be utilized to answer the research questions.

ELIGIBILITY:
Inclusion Criteria:

Maternal:

* Primary caregiver of the child with asthma seen at the community-based asthma clinic
* Female (self-identified)
* Black (self-identified)
* ≥ 18 years of age
* English-speaking
* PHQ-9 ≥ 8 during standardized screening at the child with asthma's clinic visit

Child:

* Younger than 17 years and 7 months at the date of enrollment
* Publicly insured
* Physician-diagnosed persistent asthma

Exclusion Criteria:

Maternal:

* Acutely suicidal (high risk on the C-SSRS at child's asthma clinic visit)
* Bipolar disorder or mania
* Schizophrenia
* Current substance abuse/dependence
* Current serious physical intimate partner violence (IPV)

Child:

* Significant medical co-morbidity (e.g., disorders of the cardiorespiratory system, significant developmental delay, diabetes, seizure disorder, and sickle cell disease)
* Enrolled in another intervention with a behavioral component and/or novel asthma therapeutics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identified female gender is an inclusion criterion for maternal/caregiver participation
Enrollment: 60 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Maternal depressive symptoms | T2 (3 months post-baseline)
  ≥ 50% reduction in depressive symptoms on the 9-item Patient Health Questionnaire (PHQ-9) at T2. The PHQ-9 score ranges from 0-27, with higher scores indicating more depressive symptoms. This variable will be dichotomized into 50% or greater reduction in depressive symptoms vs. less than 50% reduction in depressive symptoms from T1 to T2.

SECONDARY OUTCOMES:
Clinically significant maternal depressive symptoms | T2 (3 months post-baseline)
  9-item Patient Health Questionnaire (PHQ-9) score less than 10 (i.e., not clinically significant) at T2. The PHQ-9 score ranges from 0-27, with higher scores indicating more depressive symptoms. A score of 10 or more indicates clinically significant symptoms. This variable will be dichotomized into clinically significant and not clinically significant.
Child asthma exacerbations | T3 (6 months post-baseline)
  Number of asthma exacerbations requiring steroids in the past 6 months
Child asthma symptoms | T2 (3 months post-baseline), T3 (6 months post-baseline)
  Mother-reported number of child asthma symptom-free days during the prior 14 days
Maintenance | T3 (6 months post-baseline)
  Percentage of enrolled mothers who remain in the study
Acceptability | T2 (3 months post-baseline)
  Mean treatment satisfaction survey score on the Client Satisfaction Questionnaire
Maternal anxiety symptoms | T2 (3-months post-baseline) and T3 (6months post-baseline)
  Scores on the 7-item Generalized Anxiety Disorder sale (GAD-7). Scores range from 0-21, with higher scores indicating more anxiety.
Maternal PTSD symptoms | T2 (3 months post-baseline) and T3 (6 months post-baseline)
  Score on the PTSD Checklist for DSM-5 (PCL-5), a validated self-report measure of PTSD symptoms in adults. Scores on the PCL-5 range from 0-80, with higher scores indicating more PTSD symptoms.
Child depressive symptoms | T2 (3 months post-baseline) and T3 (6 months post-baseline)
  Mother report of child depressive symptoms on the PROMIS Parent Proxy Depressive Symptoms v3.0- Short Form 6a. Raw scores on the measure range from 6-30, with higher scores indicating more depressive symptoms.
Child anxiety symptoms | T2 (3 months post-baseline) and T3 (6 months post-baseline)
  Mother report of child anxiety symptoms on the PROMIS Parent Proxy Short Form GenPop v3.0 - Anxiety 8a. Raw scores on the measure range from 8-40, with higher scores indicating more anxiety symptoms.
Child asthma control | T2 (3 months post-baseline), T3 (6 months post-baseline)
  Dichotomized score on the Child Asthma Control Test where ACT ≥ 20 indicates controlled asthma and ACT less than 20 indicates uncontrolled asthma.
Asthma management | T2 (3 months post-baseline)
  Summary score on the Family Asthma Management System Scale (FAMSS), a clinical interview that assesses how well the family system manages the asthma of the child. The interview is recorded and rated on eight 9-point subscales that tap the various domains of asthma management, with higher scores indicating better management.
Reach | T1 (Baseline)
  The number and proportion of eligible mothers recruited into the study
Feasibility | T2 (3 months post-baseline)
  Percentage of mothers who complete at least 7 sessions of the intervention (Enhanced IPT-B)
Satisfaction | T3 (6 months post-baseline)
  Semi-structured interviews will be conducted with at least one third of Enhanced IPT-B participants to assess intervention satisfaction.
Staff-reported implementation outcomes | At the end of year 2
  Semi-structure qualitative interviews with asthma clinic staff and leadership to assess adoption, acceptability, and maintenance of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Margolis, PhD, MSW, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual and aggregate survey data (including raw and recoded data) will be shared. The data from intervention sessions with Enhanced IPT-B participants will not be shared. Summarized aggregated deidentified data from the implementation-focused process evaluation will be made available for sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The study data will be released and made available approximately 12 months following the conclusion of the award period. Datasets underlying publications will be shared at or prior to initial publication date. Data we do not publish on will be shared before the end of this award. Study data deposited in the DSDR repository will be available to the research community permanently.
Access Criteria: All shared study materials, data, and metadata will be made publicly available to researchers external to the project free of charge through the Data Sharing for Demographic Research (DSDR) digital data repository hosted by the ICPSR. The data will be findable in the DSDR repository and identifiable using a study digital object identifier provided by ICPSR.